CLINICAL TRIAL: NCT02392403
Title: Clinical Investigation of the Nucleus® CI532 Cochlear Implant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cochlear (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLTD5446
Record Dates: First submitted 2015-03-13; First posted 2015-03-19 (Estimated); Results first posted 2018-11-01 (Actual); Last update posted 2018-11-01 (Actual); Status verified 2017-07

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nucleus CI532 cochlear implant (Experimental)
  Interventions: Device: Nucleus CI532 cochlear implant

INTERVENTIONS:
Device: Nucleus CI532 cochlear implant

SUMMARY:
The aim of this study is to investigate the clinical benefit for patients implanted with the Nucleus® CI532 cochlear implant and to demonstrate the atraumatic nature of the electrode design.

Nucleus® CI532 has a pre-curved, perimodiolar array, the EA32, which is introduced into the cochlea through a straightening sheath.

ELIGIBILITY:
Inclusion Criteria:

* Eighteen years of age or older at the time of implantation
* Conventional candidate for cochlear implantation with a perimodiolar electrode array according to local criteria (excepting the exclusion criteria that follow)
* Native speaker in the local language used to assess clinical performance

Exclusion Criteria:

* Evidence of hearing loss prior to 5 years of age
* Prior cochlear implantation; i.e. having a cochlear implant in the contralateral ear, or previously implanted in either ear
* Medical or psychological conditions that contraindicate undergoing general anaesthesia or surgery
* Ossification, malformation or any other cochlear anomaly, such as common cavity, that might prevent complete insertion of the electrode array, as confirmed by medical examination
* Hearing impairment due to lesion or neuropathy of the acoustic nerve, VIII nerve or central auditory pathway
* Active middle-ear infection
* Tympanic membrane perforation
* Unrealistic expectations on the part of the subject, regarding the possible benefits, risks, and limitations that are inherent to the surgical procedure(s) and prosthetic devices
* Unwillingness or inability of the candidate to comply with all investigational requirements such as undergoing a post-operative digital volume tomography/ConeBeam scan
* Patients with existing Cerebral Spinal Fluid shunts or drains, existing perilymph fistula, skull fracture or Cerebral Spinal Fluid leak
* Patients with recurrent episodes of bacterial meningitis
* Pregnancy or breast-feeding
* Known allergies to components of the implant
* Wearing other active implants with known interference with cochlear implants

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2015-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chris J James, PhD, Study Director — Cochlear
Locations (8):
- The HEARing CRC, Melbourne, Victoria, Australia
- Service d' ORL et d'Otoneurochirurgie, CHU Toulouse Purpan, Toulouse, Midi-Pyrénées, France
- Germany (5):
  - Ear, Nose and Throat Department, University of Freiburg, Freiburg im Breisgau, Baden-Wurttemberg
  - Ear, Nose and Throat Department, Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum der J. W. Goethe-Universität Frankfurt, Frankfurt am Main, Hesse
  - Ear, Nose and Throat Department, Medizinische Hochschule, Hanover, Lower Saxony
  - Universitätsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
- Complejo Hospitalario Universitario Insular Materno Infantil, Las Palmas, Gran Canaria, Spain

REFERENCES:
- [Derived] Hey M, Wesarg T, Mewes A, Helbig S, Hornung J, Lenarz T, Briggs R, Marx M, Ramos A, Stover T, Escude B, James CJ, Aschendorff A. Objective, audiological and quality of life measures with the CI532 slim modiolar electrode. Cochlear Implants Int. 2019 Mar;20(2):80-90. doi: 10.1080/14670100.2018.1544684. Epub 2018 Nov 22. PMID 30465637

RESULTS

PARTICIPANT FLOW:
Groups:
- Nucleus CI532 Cochlear Implant: Single arm study. All participants received CI532.
Period: Overall Study
Arm/Group | Nucleus CI532 Cochlear Implant
Started | 45
Completed | 42
Not Completed | 3
Not completed — Adverse Event | 1
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 22

OUTCOME MEASURES:

1. Primary Outcome: Scalar Position of Electrode Array Determined With Computer Tomography (CT) Scan
Description: The position of the electrode array can be completely in scala tympani, completely in scala vestibuli, or may transverse from scala tympani to scala vestibuli. The position can be determined from high resolution flat panel volume tomography (Cone beam) imaging.
Time Frame: up to one month post-surgery
Population: One patient was explanted and reimplanted with a different type of device.
Measure: Count of Participants; unit: Participants
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 44
Participants
  Completely in scala tympani | 44
  Dislocation in scala vestibuli | 0

2. Secondary Outcome: Array Proximity to the Modiolus Measured Using the Wrapping Factor
Description: The ratio of the active array length and the corresponding lateral wall length
Time Frame: up to one month post-surgery
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 44
ratio | 0.62 (0.05)

3. Secondary Outcome: Surgeon Questionnaire on Implant Surgery
Description: To collect experiences using the CI532. At each surgery, the surgeon was asked whether "overall the CI532 was easy to handle and the EA32 easy to insert". We counted the number of surgeons who strongly agreed or who agreed.
Time Frame: at time of surgery
Measure: Number; unit: Surgeons
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 45
Surgeons | 38

4. Secondary Outcome: Change From Baseline in Speech Recognition in Quiet and Noise at 6 Months
Description: Change in percent correct speech recognition test scores for implant ear alone and best aided
Time Frame: baseline and 6 months post activation
Measure: Median (Inter-Quartile Range); unit: Percent correct
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 44
Percent correct
  Quiet Implant Ear | 52.500 [25.0 to 71.8]
  Quiet Best Aided | 29.668 [12.5 to 56.0]
  10 db Signal-to-Noise Ratio (SNR) Implant Ear | 63.725 [5.6 to 88.2]
  10 db Signal-to-Noise Ratio (SNR) Best Aided | 33.690 [2.5 to 63.2]

5. Secondary Outcome: Patient Reported Benefit in Health Status Assessed Via Glasgow Benefit Inventory Questionnaire
Description: The Glasgow Benefit Inventory is a single time point measure of patient reported benefit.
  A score of 0 indicates no benefit; the minimum score is -100 and the maximum is +100.
Time Frame: 6 months post activation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 42
units on a scale | 28.1 [21.577 to 34.738]

6. Secondary Outcome: Change From Baseline in Hearing Ability Assessed Via Speech Spatial Hearing Qualities Questionnaire at 6 Months
Description: Rating scale. 0=worst; 10=best
Time Frame: baseline and 6 months post activation
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 41
units on a scale | 2.22 [1.695 to 2.750]

7. Secondary Outcome: Change From Baseline in Air-conduction Pure-tone Hearing Thresholds Via an Audiogram at 6 Months
Description: We report only the change for the 500 Hz frequency.
Time Frame: baseline and 6 months post activation
Population: Note that some patients had no measurable pre-operative hearing
Measure: Median (Inter-Quartile Range); unit: Decibels
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 36
Decibels | 20 [5 to 40]

8. Secondary Outcome: Number of Adverse Events at Surgery
Time Frame: at time of surgery
Measure: Number; unit: adverse events
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 45
adverse events | 3

9. Secondary Outcome: Number of Adverse Events Post Surgery to 6 Months Post-activation
Time Frame: post surgery to 6 months post-activation
Measure: Number; unit: adverse events
Arm/Group | Nucleus CI532 Cochlear Implant
Number analyzed (Participants) | 45
adverse events | 32

ADVERSE EVENTS:
Time Frame: 16 months
Arm/Group | Nucleus CI532 Cochlear Implant
All-Cause Mortality (participants affected / at risk) | 1/45
Serious Adverse Events (participants affected / at risk) | 4/45
Other Adverse Events (participants affected / at risk) | 30/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus CI532 Cochlear Implant (N=45)
Prolonged hospitalization for re-implantation (Ear and labyrinth disorders) | 2 (2)
Death due to myocardial infarction (Cardiac disorders) | 1 (1)
Hospitalization for hysterectomy and bladder wall reinforcement (General disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nucleus CI532 Cochlear Implant (N=45)
Tinnitus (Ear and labyrinth disorders) | 7 (7)
Pain (General disorders) | 11 (11)
Dizziness and/or vertigo (Ear and labyrinth disorders) | 8 (8)
Nausea (Gastrointestinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees to send any Conference presentations/publications to the Sponsor for review at least 30 days prior to publication/presentation and after the first publication has been submitted. The Sponsor has the right to require any confidential information to be removed. If there is intellectual property disclosed, which the Sponsor intends to protect by registration such as by patent application, the Sponsor may require the release of the publication to be delayed by up to 120 days.